CLINICAL TRIAL: NCT04865874
Title: Advantages of Pulse Pressure Variation (PPV) Monitoring in Thoracic Surgery
Brief Title: GDT-PPV Protocol in Thoracic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 3901
Record Dates: First submitted 2021-04-14; First posted 2021-04-29 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Thoracic Surgery; Fluid-therapy
Keywords: pulse pressure variation; zero balance; single-lung ventilation

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PPV-GDT (Experimental): Intra-operative fluid-therapy based (lactated Ringer) on continous PPV monitoring (target ≤5.8%)
  Interventions: Other: PPV-GDT
- Zero balance (Active Comparator): Intra-operative fluid-therapy (lactated Ringer) based on 1:1 compensation of urinary output
  Interventions: Other: Zero-balance

INTERVENTIONS:
Other: PPV-GDT — fluid-therapy based on PPV monitoring
  Arms: PPV-GDT
Other: Zero-balance — fluid-therapy based on urinary output balance
  Arms: Zero balance

SUMMARY:
Peri-operative fluid-therapy is extremely important in thoracic surgery, because excessive administration of fluids during one-lung ventilation is correlated to an increasing risk of postoperative respiratory complications.

Therefore, current guidelines on peri-operative management of patients undergoing thoracic surgery suggest a conservative fluid management strategy, based on intra-operative fluid loss replacement and maintenance of euvolemia.

Nevertheless, intra-operative fluid loss estimation and consequently the correct infusion rate adoption are quite difficult to be addressed in clinical practice, and this often prevents the euvolemia maintenance in the peri-operative period.

This limit claims the necessity to adopt new methods of fluid-therapy administration in thoracic surgery; among these the most promising is the "Goal-Directed Therapy" (GDT). GDT protocols based on Stroke Volume Variation (SVV) or Pulse Pressure Variation (PPV) monitoring have been adopted successfully in major and cardiac surgery but not yet in thoracic surgery.

The aim of this randomized study is to evaluate the effects of a PPV-GDT fluid management protocol versus a conservative "zero-balance" protocol on intrapulmonary gas exchanges, in patients undergoing single-lung ventilation during thoracic surgery.

DETAILED DESCRIPTION:
The intra-operative fluid-therapy (using lactated Ringer) will be based on pulse pressure variation (PPV group) with a target ≤5.8% or on compensation (1:1) of urine output (zero balance group).

In both groups an intraoperative background infusion of lactated Ringer at 1-2 ml/kg/h will be administered.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients scheduled for Video-assisted thoracic surgery (VATS) lobectomy

Exclusion Criteria:

* Patients who will not sign the informed consent
* Obesity (BMI > 35 kg/m2)
* Cardiovascular disease (heart failure, arrhythmia)
* OSAS requiring or not C-PAP therapy
* Chronic alcoholism
* intraoperative blod loss> 1500 ml
* One-lung ventilation duration< 60 min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2021-09-21 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
PaO2/FiO2 ratio | 15 minutes after extubation
  Ratio of arterial oxygen partial pressure (PaO2 in mmHg) to fraction of inspired oxygen (FiO2)

SECONDARY OUTCOMES:
Postoperative pulmonary complications | Up to 3 days after surgery
  e.g. Atelectasis, pneumonia, lung edema, pleural effusion, hypoxemia
In-hospital stay | Days until discharge, an average of 5 days
  Hospital stay duration

CONTACTS AND LOCATIONS:
Overall Officials: Paola Aceto, MD,PhD, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- UOC Anestesia delle Chirurgie Generali e dei Trapianti, Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Lazio/Rome, Italy

IPD SHARING:
Plan to Share IPD: No